CLINICAL TRIAL: NCT06633250
Title: Effect of a Hydrolyzed Rice Protein-based Formula on Growth, Tolerance, and Health-related Quality of Life in Infants With Cow's Milk Protein Allergy: a Randomized Nutritional Clinical Study
Brief Title: Effect of a Hydrolyzed Rice Protein-based Formula on Growth, Tolerance, and Health-related Quality of Life in Infants With Cow's Milk Protein Allergy.
Acronym: RIGHT-GO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2204INF
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cow Milk Protein Allergy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Formula (Experimental): Hydrolyzed rice protein formula
  Interventions: Other: Test Formula
- Control Formula (Active Comparator): Commercially available extensively hydrolyzed cow's milk formula
  Interventions: Other: Control Formula

INTERVENTIONS:
Other: Test Formula — Hydrolyzed rice protein formula
  Arms: Test Formula
Other: Control Formula — Commercially available extensively hydrolyzed cow's milk formula
  Arms: Control Formula

SUMMARY:
The main purpose of this study is to demonstrate that the growth of infants fed with the Test Formula is non-inferior those fed with the Control Formula. The study will also evaluate the gastrointestinal tolerance, quatliy of life and acceptability of the new rice protein-based formula in infants with cow's milk protein allergy (CMPA).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained from at least one parent (or legally acceptable representative [LAR]), if applicable)
2. Infant gestational age ≥ 37 completed weeks
3. Infant birth weight of ≥ 2.5 kg and ≤ 4.5 kg
4. Singleton birth
5. Infant age ≤ 8 months
6. Mother has previously decided to fully formula-feed, and infant is no longer breastfeeding or receiving breast milk
7. Suspected CMPA as per standard clinical practice and in conjunction with at least 2 symptoms present from the list shown below:

   1. Inconsolable crying, regurgitation, liquid stools or constipation, skin atopic lesion, cow's milk provoked temporary urticaria/angioedema or vomiting, bloody streaks in stool, or respiratory symptoms
   2. For diagnosis based on either a positive IgE blood test, skin prick test or food challenge, only at least 1 symptom from above list needs to be present
8. Infant is receiving a strict cow's milk elimination diet and will continue receiving this diet until the completion of the study
9. Infant's parent(s)/LAR is of legal age of majority, must have parental authority, must understand the informed consent form and other study documents, and is willing and able to fulfill the requirements of the study protocol

Exclusion Criteria:

1. History of intolerance to eHF formula
2. Any chronic medical diseases (except atopic eczema), chromosomal or major congenital anomalies (based on medical history and/or commonly performed diagnostic criteria)
3. Major gastrointestinal disease / abnormalities (other than CMPA)
4. Known or suspected lactose intolerance or malabsorption
5. Known or suspected soy allergy
6. Glucose-galactose malabsorption
7. Rice protein allergy or intolerance (e.g., rice protein-induced enterocolitis syndrome).
8. Immunodeficiency
9. Persistent wheeze or chronic respiratory disease
10. Severe uncontrolled eczema
11. History of severe anaphylactic reaction (e.g., requiring ≥ 2 doses of epinephrine) to cow's milk or breast milk at any time prior to enrollment
12. Weight-for-age value < -2 or > 2 standard deviations from the WHO Child Growth Standards median at enrollment
13. Height-for-age < -2 or > 2 standard deviations from the WHO Child Growth Standards median at enrollment
14. Infant's parent has other medical or psychiatric condition that, in the judgement of the investigator, would make the infant inappropriate for entry into the study
15. Currently participating or having participated in another interventional clinical study within 4 weeks prior to enrollment

Max Age: 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Weight-for-age z-score at 4 months post-enrollment | From enrollment to 4 months post-enrollment
  Weight measured in g and expressed in z scores according to the World Health Organization (WHO) Child Growth Standards.

SECONDARY OUTCOMES:
Weight | Monthly from enrollment to 4 months post-enrollment
  Weight (g and z-scores)
Length | Monthly from enrollment to 4 months post-enrollment
  Length (cm and z-scores)
Head circumference | At enrollmentn and 4 months post-enrollment
  Head circumference (cm and z-scores)
Tibia lenght | At enrollmentn and 4 months post-enrollment
  Tibia (cm)
Femur lenght | At enrollmentn and 4 months post-enrollment
  Femur (cm)
Gastrointestinal Symptoms | Monthly from enrollment to 4 months post-enrollment, and 7 days after enrollment
  The Infant Gastrointestinal Symptom Questionnaire (IGSQ) will be used to assess GI tolerance. The IGSQ is a validated instrument that includes 13 questions in 5 domains (stooling, spitting-up/vomiting, crying, fussiness, and flatulence) and total scores range from 13 (best) to 65 (worst) for overall GI symptom burden.
Gastrointestinal Symptoms | First 7 days post enrollment
  A daily GI tolerance questionnaire will be used.
Stool frequency and consistency | At enrollment
  A retrospective 1-day stool record including the Brussels Infant and Toddler Stool Scale will be used.
Stool frequency and consistency | 2 months and 4 months post-enrollment
  A 3-day stool diary including the Brussels Infant and Toddler Stool Scale will be used.
Cow's Milk-related Allergy Symptom | Monthly from enrollment to 4 months post-enrollment
  The Cow's Milk-related Symptom Score (CoMiSS) will be used to assess symptoms related to CMPA. The CoMiSS questionnaire contains 6 items and generates a score based on gastrointestinal, dermatological, respiratory, and general symptoms (total score range 0-33), which may be associated with CMPA .
Food Allergy Quality of Life | At enrollment and 4 months post-enrollment
  The Food Allergy Quality of Life Questionnaire (FAQLQ-PF) will be used. It is a validated instrument with 30 items in 3 domains (emotional impact, food-related anxiety, dietary and social restrictions).
Parental self-efficacy in managing food allergy | At enrollment and 4 months post-enrollment
  Parental self-efficacy in managing their child's food allergy will be assessed using the Food Allergy Self-Efficacy Scale for Parents (FASE-P). The FASE-P is a validated instrument with 21 items.
Parent-reported infant health-related quality of life | At enrollment and 4 months post-enrollment
  Parent-reported infant health-related quality of life will be assessed using the Infant and Toddler Quality of Life Questionnaire - Short Form (ITQOL-SF47). The ITQOL-SF47 is a validated instrument with 47 items.
Complementary food intake | At enrollment, 2 months post-enrollment and 4 months post-enrollment
  Total energy and macronutrient intake calculated from food recalls / diaries.
Formula compliance | Monthly from enrollment to 4 months post-enrollment
  A questionnaire will be used to assess formula compliance.
Formula liking | 4 months post-enrollment
  A questionnaire will be used to assess formula liking.
Safety - Occurence of AE | From enrollment to 4 months post-enrollment
  Adverse Events will be collected.

CONTACTS AND LOCATIONS:
Locations (19):
- Charité Universitätsmedizin Berlin, Berlin, Germany
- Italy (5):
  - Azienda Ospedaliera Universitaria Federico II, Naples
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - AOUP Ospedale Santa Chiara, Pisa
  - Ospedale Pediatrico Bambino Gesu, Rome
  - AO Ordine Mauriziano, Turin
- Poland (13):
  - Poliklinika Ginekologiczno-Położnicza Arciszewscy, Bialystok
  - Centrum Medyczne Pratia, Bydgoszcz
  - IN-VIVO Bydgoszcz, Bydgoszcz
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny, Bydgoszcz
  - Vitamed Galaj i Cichomski, Bydgoszcz
  - BioMedical Centers, Janki
  - Centrum Medyczne Plejady, Krakow
  - Jagiellonian University Medical College, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Lodz
  - ETG Lublin, Lublin
  - Korczowski Bartosz Gabinet Lekarski, Rzeszów
  - Alergo-Med Specjalistyczna Przychodnia Lekarska, Tarnów
  - University Hospital of Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: No